CLINICAL TRIAL: NCT00483600
Title: Studies of Fondaparinux in Patients With Renal Dysfunction: PK Study of Fondaparinux in Outpatients With Renal Dysfunction
Brief Title: Pharmacokinetic Study of Fondaparinux in Outpatients With Renal Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00001571
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-02

CONDITIONS: Kidney Diseases
Keywords: Fondaparinux; Pharmacokinetic
MeSH Terms: conditions — Kidney Diseases | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- no arms/one group (Experimental)
  Interventions: Drug: fondaparinux

INTERVENTIONS:
Drug: fondaparinux — injections of 2.5mg every other day for 4 weeks
  Other Names: Arixtra

SUMMARY:
To determine the appropriate dose and safety of a preventative dose of fondaparinux, an anticoagulant medication (blood thinner) in patients with kidney disease.

DETAILED DESCRIPTION:
This study will evaluate the PK of fondaparinux in patients who have renal insufficiency. Fondaparinux is cleared from the body mainly by the kidneys. Therefore in patients with kidney diseases, full doses of fondaparinux could cause bleeding problems. The correct dose of fondaparinux that should be used in patients with kidney disease is not known. The purpose of this research is to determine the PK and safety of a preventative dose (2.5mg subcutaneously every other day) of fondaparinux for patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients in the Medicine and Nephrology clinics who are 18 years or older,
* Outpatients in the Medicine and Nephrology clinics who have an estimated creatinine clearances between 20-30ml/min,
* Outpatients in the Medicine and Nephrology clinics who are able to give consent will be included.

Exclusion Criteria:

* anticoagulation therapy for thrombosis or other indication
* pregnant or breast-feeding
* hypersensitivity to fondaparinux
* subjects also will be excluded if there is concern for an increased risk of bleeding which includes the following:

  * known bleeding disorder (see Section 8. Hemostatic Assessment)
  * blood transfusion in the past 3 months
  * acute ulcer disease with past 3 months
  * platelet count < 120,000 mm3
  * prolonged baseline prothrombin time (PT) or activated partial thromboplastin time (aPTT) above upper limit of normal laboratory range
  * major trauma or surgery within two weeks prior to enrollment
  * history of intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
PK parameters (half-life, area-under-the curve, and peak serum concentration) | after day 7 and after day 27

SECONDARY OUTCOMES:
Anti-factor Xa levels and assessment for bleeding(complete blood count) | days 3, 13 and 19

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Ortel, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States